CLINICAL TRIAL: NCT04913662
Title: Safety of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Using Paclitaxel in Gastric Cancer Patients With Peritoneal Metastasis
Brief Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Using Paclitaxel in Gastric Cancer Patients With Peritoneal Metastasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Hospicare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH_PIPAC_PTX
Record Dates: First submitted 2021-04-26; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Stomach Neoplasm; Peritoneal Metastases
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PIPAC Paclitaxel with FOLFOX (Experimental): PIPAC (Paclitaxel) + Systemic mFOLFOX6(5-FU, Oxaliplatin, Leucovorin)
  Interventions: Procedure: Pressurized Intraperitoneal Aerosol Chemotherapy

INTERVENTIONS:
Procedure: Pressurized Intraperitoneal Aerosol Chemotherapy — Aerosolization of chemotherapic agent for intraperitoneal chemotherapy

SUMMARY:
This is a phase I trial investigating the safety of pressurized intraperitoneal aerosol chemotherapy (PIPAC) using paclitaxel combined with intravenous FOLFOX therapy for gastric cancer patients with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as gastric adenocarcinoma
* Imaging scans or diagnostic laparoscopic findings suggestive of peritoneal metastasis
* HER-2 negative tumor
* Laboratory tests adequate for chemotherapy (within 2 weeks of enrollment)
* Absolute Neutrophil Count: ≧ 1,500/mm³
* Hemoglobin level: ≧ 8.0g/dL
* Platelet Count: ≧ 10×104/mm³
* AST (GOT), ALT (GPT): ≦ 100U/L
* Total Bilirubin: ≦ 2.0mg/dL
* Creatinine Clearance (CCl): ≧ 50mL/min
* ECOG 0 - 2

Exclusion Criteria:

* Patients with other major medical disease or malignant tumors other than gastric cancer
* Contraindication to 5-FU, Oxaliplatin, Leukovorin or Paclitaxel
* Pregnant, breast-feeding women or with birth plan
* History of gastrointestinal surgery
* Patients refusing treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-04-26 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Recommended dose | Dose-limiting toxicity within 2 weeks after 1st intraoperative PIPAC (each cycle is 6 weeks)
  Recommended dose of paclitaxel for a phase II trial

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR